CLINICAL TRIAL: NCT02289378
Title: Dose-dense Biweekly Docetaxel, Oxaliplatin and 5-fluorouracil as First-line Treatment in Advanced Gastric Cancer
Acronym: DaeMon-Plus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lan Ping, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DaeMon Plus
Record Dates: First submitted 2014-11-07; First posted 2014-11-13 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Docetaxel, Oxaliplatin and Fluorouracil
MeSH Terms: interventions — Docetaxel; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel, Oxaliplatin and 5-Fu (Experimental): Docetaxel 50mg/m2 Oxaliplatin 85mg/m2 5-Fu 2800mg/m2 Repeated every two weeks
  Interventions: Drug: Docetaxel, Oxaliplatin and 5-Fu

INTERVENTIONS:
Drug: Docetaxel, Oxaliplatin and 5-Fu — To investigate the triplet regimen in the first-line therapy of advanced chemotherapy

SUMMARY:
This is an open-label, phase II study to evaluate the efficacy and safety of biweekly docetaxel, Oxaliplatin and de Gramont regimen on unresectable gastric adenocarcinoma in the first-line therapy.

DETAILED DESCRIPTION:
Docetaxel 50mg/m2 Oxaliplatin 85mg/m2 5-Fu 2800mg/m2 Repeated every two weeks

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Patients with histologically or cytologically confirmed unresectable gastric adenocarcinoma whose ECOG performance status are 0-2
* Presence of measurable disease by radiographic study (including CT or MRI scan, or chest x-ray) or physical examination
* At least 3 weeks since last major surgery
* At least 12 months since last adjuvant chemotherapy
* At least 6 weeks since prior radiotherapy providing that the extent and site of radiotherapy fields are such that marked bone marrow suppression is NOT expected
* Patients who have received palliative radiotherapy must have recovered from any reversible toxic effects e.g. nausea and vomiting caused by radiation of fields
* Patients with reproductive potential must use effective BC
* Required Screening Laboratory Criteria:

Hemoglobin 90g/L WBC 3.5 x 109/L Neutrophils 1.5 x 109/L Platelets 100 x 109/L Creatinine 133 umol/L and creatinine clearance 60 mL/min

* A probable life expectancy of at least 6 months

Exclusion Criteria:

* Brain metastases
* Female of childbearing potential, pregnancy test is positive
* Concomitant malignancies or previous malignancies other than gastric cancer within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or low grade prostate cancer
* Active infection
* Concurrent severe medical problems unrelated to the malignancy, which would significantly limit full compliance with the study or expose the patient to extreme risk
* Sexually active patients refusing to practice adequate contraception; Patients with conditions which might affect absorption of an oral drug (for example intermittent obstruction) unless discussed and agreed with principal investigator
* History of grade 3 or 4 toxicity to fluoropyrimidines

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years

SECONDARY OUTCOMES:
Response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ping Lan, MD, Study Chair — The Sixth Affilated Hospital of Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China